CLINICAL TRIAL: NCT03679494
Title: Effectiveness of Implementing Shared Decision-Making on Quality of Care Among Patients With Lumbar Degenerative Diseases: A Cluster Randomized Controlled Trail
Brief Title: Effectiveness of Implementing Shared Decision-Making on Quality of Care Among Patients With Lumbar Degenerative Diseases.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: N201712035
Record Dates: First submitted 2018-09-06; First posted 2018-09-20 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-12

CONDITIONS: Lumbar Degenerative Disease; Shared Decision Making; Patient Decision Aids; Evidence-based Medicine; Quality of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDM intervention group (Experimental): Using shared decision making support tool for intervention
  Interventions: Other: Shared decision making support tool
- Usual care group (No Intervention): No intervention, just continue using usual care

INTERVENTIONS:
Other: Shared decision making support tool — Health education materials containing treatments and questions about patient values to help patients make the most appropriate decisions
  Arms: SDM intervention group

SUMMARY:
Background:

Shared decision making (SDM) is a patient-centered and evidence-based model of clinical decision making. The feature of SDM is that clinicians work together with patients to plan the most appropriate and practical treatment for patients based on the patients' preferences and values. Recently, SDM has been implemented throughout the world to improve patients' health literacy and to have a better understanding of the treatment options, thereby improving patient-doctor communication and promoting the quality of care.

Lumbar degenerative disease is a critical public health issue in the aging society. SDM now becomes an important process because there is no consensus of evidence-based practice guidelines among the multiple complex treatment options for patients with lumbar degenerative disease. In addition, there is a lack of evidence to support the effect of patient decision aids (PDAs) to promote the quality of healthcare for patients with lumbar degenerative disease in Taiwan.

Purposes:

This project has two purposes. The first purpose is to develop a multimedia interactive patient doctor communication system called the Taiwan Shared Decision Making for Lumbar Spine Treatment (Taiwan SDM LumST). The second and ultimate purpose is to conduct a cluster randomized controlled trial (cRCT) for the validation of the integrated SDM model and the effectiveness of SDM related outcome indicators.

Methods:

In the first year of the 3-year project, investigators will develop the SDM communication teaching materials, PDAs, as well as the computerized platform of Taiwan SDM LumST through focus groups and consensus meetings. In the second to third year, investigators will recruit 130 patients with lumbar degenerative disease to participate in double blind cRCT in the affiliated hospitals of Taipei Medical University. Investigators will use structural equation modeling to validate the factors of the SDM model and adopt generalized linear regression models with generalized estimating equations to examine the immediate, short-term, and long-term benefits of the Taiwan SDM LumST in implementing the SDM model among patients with lumbar degenerative disease.

Expected results:

Investigators expect that the implementation of the Taiwan SDM LumST system will significantly improve the patients' decision preference, health literacy in the care of lumbar degenerative disease, and self-efficacy in SDM. It will also promote the health care quality and health outcomes (e.g., participation in SDM, quality of decisions, regret in decisions, health outcomes, and quality-of-life) in patients with lumbar degenerative disease.

Expected impacts on the society, economy, and academic developments:

The Taiwan SDM LumST will be an efficient and effective way to facilitate patient doctor communication and thereby, promote health outcomes and improve the quality of decisions made by patients with lumbar degenerative disease. No computerized interactive PDA of SDM system for patients with lumbar degenerative disease exists in Taiwan yet. Thus, our system would be the first in Taiwan for the lumbar degenerative population. Investigators hope that the Taiwan SDM LumST will not only contribute to academic research, but also facilitate SDM between patients and healthcare professionals in order to improve patient safety and enhance the quality of care in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* First-time diagnosis of Spine Degeneration Diseases ICD-10 codes M48.05-08, M43.05-08, M43.15-18, M54.5; ICD-9 codes 724.01-02、724.09、724.2、738.4
* Ability to follow instructions and complete the interviews
* Age>20 years
* Interested to participate and able to sign consent

Exclusion Criteria:

* Cognitive impairment (Mini-Mental State Examination scores<24)
* Having major mental diseases (i.e., depression, dementia, delirium, etc.)
* Inability to read/answer questionnaires

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2019-12-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SDM Intervention Group: Using shared decision making support tool for intervention
  Shared deicision making support tool: Health education materials containing treatments and questions about patient values to help patients make the most appropriate decisions
Period: Overall Study
Arm/Group | SDM Intervention Group | Usual Care Group
Started | 67 | 63
Completed | 67 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SDM Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Continuous [Median (Standard Deviation); unit: years] | 56.46 (14.853) | 55.78 (15.315) | 56.13 (15.024)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 38 | 83
  Male | 22 | 25 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 67 | 63 | 130
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Change of Patients' Control Preference
Description: Use Control Preference Scale to measure the patients' preferred role whether change in making decisions with the medical provider before intervention and after intervention. It consists of five cards, each of which presents a different character in medical decision-making in a cartoon pattern, and performs a series of comparisons to rank the preference.
Time Frame: Before intervention, up to 12 weeks after intervention
Population: Patients lost after 12 weeks of intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | SDM Intervention Group | Usual Care Group
Number analyzed (Participants) | 67 | 62
Participants
  Before intervention: Make final selection I will receive | 1 | 1
  Before intervention: Make selection with doctor's opinion | 16 | 14
  Before intervention: Make selection with doctor | 38 | 35
  Before intervention: Make selection by doctor | 12 | 12
  Up to 12 weeks after intervention: number analyzed (Participants) | 56 | 57
  Up to 12 weeks after intervention: Make final selection I will receive | 0 | 3
  Up to 12 weeks after intervention: Make selection with doctor's opinion | 1 | 0
  Up to 12 weeks after intervention: Make selection with doctor | 52 | 51
  Up to 12 weeks after intervention: Make selection by doctor | 3 | 3

2. Primary Outcome: The Change of Patients' Decision Self-efficacy
Description: Use Decision Self Efficacy Scale to measure patients' self-confidence and belief in measuring the ability of patients to participate in decision-making. It has 11 items with 5 level Likert scale. The scale range is 0-100, higher scores indicate better decision self-efficacy.
Time Frame: Before intervention, after intervention immediately, up to 12 weeks after intervention
Population: Patients lost after the intervention immediately and up to 12 weeks after intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SDM Intervention Group | Usual Care Group
Number analyzed (Participants) | 67 | 62
score on a scale
  Before intervention | 77.78 (16.78) | 79.51 (19.31)
  After intervention immediately: number analyzed (Participants) | 66 | 62
  After intervention immediately | 88.57 (10.03) | 81.27 (18.96)
  Up to 12 weeks after intervention: number analyzed (Participants) | 56 | 57
  Up to 12 weeks after intervention | 84.01 (18.61) | 85.39 (16.91)

3. Secondary Outcome: Assess Decision Process Quality in Making the Decision
Description: Assess whether the medical personnel have sufficiently communicated with patients when making the decision by 9-item Shared Decision Making Questionnaire(SDM-Q-9). It has 9 items and is divided into 0 to 5 scores, 0 points = very disagree, 1 point = roughly disagree, 2 points = partial disagreement, 3 points = partial consent, 4 points = roughly agree, 5 points = very agree. After the total score of each question is added, the initial total score is 0 to 45 points. Divide the initial total score by 9 and multiply by 20 to get the final score from 0 to 100. The higher the score means the better the decision-sharing on behalf of the patient.
Time Frame: After intervention immediately
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SDM Intervention Group | Usual Care Group
Number analyzed (Participants) | 66 | 62
score on a scale | 87.47 (12.30) | 81.76 (19.55)

4. Secondary Outcome: Assess Patients' Satisfaction With Decision
Description: Use Satisfaction with Decision Scale to assess patients satisfaction with health care decisions. It has 6 items with 5 level Likert scale. 1 point = very disagree, 2 points = disagree, 3 points = disagree or disagree, 4 points = agree, 5 points = very agree. After the total score of each question is added, the initial total score is 6 to 30 points. The higher the score, patients are more satisfied with the decision.
Time Frame: After intervention immediately, up to 12 weeks after the intervention
Population: The patients lost up to 12 weeks after the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SDM Intervention Group | Usual Care Group
Number analyzed (Participants) | 66 | 62
score on a scale
  After intervention immediately | 26.29 (3.40) | 25.06 (4.60)
  Up to 12 weeks after the intervention: number analyzed (Participants) | 56 | 57
  Up to 12 weeks after the intervention | 26.02 (3.89) | 25.44 (4.71)

5. Secondary Outcome: Assess Patients' Decisional Conflict
Description: Use the Decisional Conflict Scale to assess patients whether have a conflict or something not sure about making the decision. It has 16 items with 5 levels Likert scale. 0 points = yes, 1 point = about yes, 2 points = uncertainty, 3 points = probably not, 4 points = no. After the total score of each question is added, the initial total score is 0 to 64 points. Divide the initial total score by 16 and multiply by 25 to get the final score from 0 to 100. The higher the score, patients have more conflict with the decision.
Time Frame: After intervention immediately and up to 12 weeks after intervention
Population: Patients lost after up to 12 weeks after intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SDM Intervention Group | Usual Care Group
Number analyzed (Participants) | 66 | 62
score on a scale
  After intervention immediately | 10.30 (10.46) | 18.25 (18.44)
  Up to 12 weeks after intervention: number analyzed (Participants) | 56 | 57
  Up to 12 weeks after intervention | 15.77 (17.56) | 15.27 (14.75)

6. Secondary Outcome: Assess the Degree of Disability of Lower Back Pain
Description: Use the Oswestry Disability Index to measure lower back pain patients' degree of disability. It has 10 items (Pain, self-care, bring, walking, sitting, standing, sleeping, sex, social, travelling). After adding up the total score of each item, the initial total score is 0 to 50 points. Then divide the total score by 5 and multiply by 20 to get the final score of 0 to 100. Higher scores indicate a more severe disability.
Time Frame: Before intervention, up to 12 weeks after intervention
Population: Patients lost up to 12 weeks after intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SDM Intervention Group | Usual Care Group
Number analyzed (Participants) | 67 | 62
score on a scale
  Before intervention | 24.38 (15.67) | 24.62 (12.90)
  Up to 12 weeks after intervention: number analyzed (Participants) | 55 | 57
  Up to 12 weeks after intervention | 24.22 (31.06) | 21.12 (25.20)

7. Secondary Outcome: Assess the Quality of Healthy Living About Patients
Description: Use the EQ-5D-5L scale to measure patients' quality of healthy living. It has 5 items (Mobility, Self-care, Usual activities, Pain/discomfort, Depression/anxiety). Each item contains 5 levels: 1= no difficulty, 2= slight difficulty, 3= moderate difficulty, 4= serious difficulty, 5= extremely serious difficulty. The higher the score has the worse the health. Then, the score calculation of the European Five-Dimensional Health Scale is based on the calculation formula published by the EuroQol Group. Based on 5 combinations of different severity levels, a score of 0 to 1 is obtained. 0 is the least healthy and 1 is the most healthy.
Time Frame: Before intervention, up to 12 weeks after intervention
Population: Patients lost up to 12 weeks after intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SDM Intervention Group | Usual Care Group
Number analyzed (Participants) | 67 | 62
score on a scale
  Before intervention | 0.70 (0.17) | 0.72 (0.13)
  Up to 12 weeks after intervention: number analyzed (Participants) | 55 | 57
  Up to 12 weeks after intervention | 0.86 (0.17) | 0.85 (0.18)

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: This is a questionnaire interview study, if patients are tired or feel unwell due to the long questionnaire, they can stop the visit at any time and immediately contact the relevant medical unit.
Arm/Group | SDM Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/63
Other Adverse Events (participants affected / at risk) | 0/67 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT03679494/Prot_SAP_000.pdf